CLINICAL TRIAL: NCT01287156
Title: Evaluation and Diagnosis of Potential Research Subjects With Traumatic Brain Injury (TBI)
Brief Title: Evaluation and Diagnosis of Potential Research Subjects With Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Center for Neuroscience and Regenerative Medicine (CNRM) (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110084; 11-N-0084
Record Dates: First submitted 2011-01-29; First posted 2011-02-01 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2026-01-06

CONDITIONS: Traumatic Brain Injury
Keywords: Recruitment; TBI; Screening; Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Subjects with diagnosed or suspected TBI or postconcussive syndrome

SUMMARY:
Background:

- The Center for Neuroscience and Regenerative Medicine is working to improve physicians' understanding of brain injury. More information is needed on traumatic brain injury (TBI), especially how well a person recovers from TBI and how the brain changes over time in people with TBI. To conduct this research, the center is sponsoring a number of research studies on TBI and is interested in evaluating individuals with TBI or post-concussive syndrome to determine if they might be eligible for future studies.

Objectives:

- To develop a pool of individuals with traumatic brain injury and post-concussive syndrome for future research studies.

Eligibility:

- Individuals at least 18 years of age who have symptoms of or have been diagnosed with traumatic brain injury or post-concussive syndrome and are willing to participate in future studies.

Design:

* Participants will be screened with an initial telephone interview, and will be asked to come to the National Institutes of Health for an in-person screening visit.
* At the screening visit, participants will provide a medical history, have a physical examination and complete a study questionnaire on their TBI and its symptoms, including how the injury occurred, when it occurred, and any previous brain-related injuries.
* Subjects may also return for a second visit at the NIH CC if eligible.
* Each visit may involve blood samples, an MRI scan, and a series of tests to evaluate brain function.
* Participants will also provide contact information to enable researchers to contact them for future studies.

DETAILED DESCRIPTION:
Objective

This screening and registry protocol is designed to facilitate subject recruitment for the Center for Neuroscience and Regenerative Medicine (CNRM) sponsored clinical research studies on traumatic brain injury (TBI) at the National Institutes of Health (NIH) and participating CNRM sites. This protocol will serve as a first step for evaluating subjects for possible inclusion in CNRM sponsored natural history, observational, or interventional protocols. Other approved CNRM protocols may continue to recruit subjects directly into their respective studies, and may refer subjects to this study.

The objective of this protocol is to develop a subject recruitment database that will house preliminary data on research subjects who are interested in and potentially eligible for current and future CNRM sponsored protocols. The effectiveness of the recruitment methods utilized in this protocol will be evaluated to determine the most successful outreach approaches and recruitment tools for the enrollment of TBI or post concussive study subjects.

Study Population

This protocol will enroll 2500 male and female adult subjects with signs/symptoms or diagnosis of TBI or post-concussive syndrome, from participating sites, other CNRM sponsored protocols and within the community using various methods of outreach and advertisement.

Design

This study involves an initial study visit conducted in one of two ways: at the NIH Clinical Center,or at the participating site. Subjects enrolled acutely and/or at a participating site may also be provided the option to complete an additional visit at the NIH CC after their initial visit. Based on the information obtained during the initial study visit, the subject will be referred to appropriate CNRM protocols for further protocol-specific screening prior to enrollment, or informed that s/he is not eligible for any other actively enrolling CNRM studies at this time. Study procedures may include: physical exam, medical history, nursing evaluation, questionnaires completed by interview, blood and urine sample collection, and magnetic resonance imaging (MRI).

Follow-up visits will be conducted by telephone at regular intervals for a year, and then ad hoc at potential referral eligibility to update contact information and collect outcome data. No treatment is offered under this protocol.

Outcome Measures

The outcome measures include accrual of subjects, retention of enrolled subjects and loss to follow-up, and referral number and rate of enrolled subjects to other CNRM studies. In addition, we will evaluate the frequency and certainty of injury classification (possible, probable, or definite TBI).

ELIGIBILITY:
* INCLUSION CRITERIA:

To be included, participants must meet all of the following:

* Age greater than or equal to 18 years of age
* Report having symptoms or diagnosis of concussion, TBI, post concussional syndrome, or post concussional disorder.
* Are able to provide informed consent or, have a legally authorized representative (LAR) provide consent.
* Are willing to have their contact information and data shared and stored by the CNRM for referral to current and future CNRM studies

EXCLUSION CRITERIA:

-Are unwilling or unable to cooperate with the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrollment in this protocol will occur at a participating site MedStar Washington Hospital Center (WHC) or Johns Hopkins Suburban Hospital (Suburban), or at the NIH Clinical Center (NIH CC). Applicable study procedures will depend on the visit site, diagnostic certainty, and logistic considerations such as distance from NIH and feasibility of transport. All subjects will undergo a study visit at a participating enrollment site and/or the NIH Clinical Center. Subjects enrolled acutely at the NIH CC may undergo an additional study visit at the NIH. Phone follow-up will occur at 6-months, 1 year from initial consent. Additional subject follow-up contact will be made should @@@a subject become eligible for referral to another eligible protocol.@@@
Sampling Method: Non-Probability Sample
Enrollment: 1328 (Actual)
Dates: Start 2013-01-10 (Actual)

PRIMARY OUTCOMES:
Develop a patient recruitment database. | intermittently
  To facilitate patient recruitment to CNRM sponsored TBI related clinical research at the NIH and participating CNRM sites by developing a patient recruitment database.

SECONDARY OUTCOMES:
To evaluate the effectiveness of the recruitment methods utilized in this protocol and determine the most successful outreach approaches and recruitment tools for the recruitment and enrollment of TBI study participants | Annually, or as needed ad hoc

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence L Latour, Ph.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (4):
- United States (4):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Suburban Hospital, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Virginia Commonwealth University Medical Center, Richmond, Virginia

REFERENCES:
- [Background] Rutland-Brown W, Langlois JA, Thomas KE, Xi YL. Incidence of traumatic brain injury in the United States, 2003. J Head Trauma Rehabil. 2006 Nov-Dec;21(6):544-8. doi: 10.1097/00001199-200611000-00009. PMID 17122685
- [Background] Langlois JA, Rutland-Brown W, Wald MM. The epidemiology and impact of traumatic brain injury: a brief overview. J Head Trauma Rehabil. 2006 Sep-Oct;21(5):375-8. doi: 10.1097/00001199-200609000-00001. PMID 16983222
- [Background] Kraus MF, Smith GS, Butters M, Donnell AJ, Dixon E, Yilong C, Marion D. Effects of the dopaminergic agent and NMDA receptor antagonist amantadine on cognitive function, cerebral glucose metabolism and D2 receptor availability in chronic traumatic brain injury: a study using positron emission tomography (PET). Brain Inj. 2005 Jul;19(7):471-9. doi: 10.1080/02699050400025059. PMID 16134735
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-N-0084.html